CLINICAL TRIAL: NCT02396771
Title: Effect of Uterine Massage Versus Sustained Uterine Compression on Blood Loss and Maternal Pain After Vaginal Delivery: a Randomized Controlled Trial
Brief Title: Effect of Uterine Massage Versus Sustained Uterine Compression on Blood Loss After Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Labib Ghulmiyyah, Associate Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OGY.LG.02
Record Dates: First submitted 2015-03-19; First posted 2015-03-24 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine; Massage; Compression
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Massage (Experimental): Women allocated to the uterine massage group will be provided with 2 minutes of trans-abdominal uterine massage starting promptly after placental delivery.
  Interventions: Procedure: Uterine Massage
- Compression (Experimental): Women allocated to the uterine compression group will be provided with 2 minutes of sustained trans-abdominal uterine compression starting promptly after placental delivery.
  Interventions: Procedure: Uterine Compression

INTERVENTIONS:
Procedure: Uterine Massage — The massage will be performed as follows: palpating the uterine fundus, manually stimulating the fundus and the whole body of the uterus using fingers and palms steadily and repetitively.
  Arms: Massage
Procedure: Uterine Compression — The sustained uterine compression will be performed as follows: placing one hand in the vagina and pushing against the body of the uterus while the other hand compresses the fundus from above through the abdominal wall.
  Arms: Compression

SUMMARY:
The purpose of this study is to compare trans-abdominal uterine massage to sustained uterine compression after vaginal delivery with respect to blood loss and maternal pain. It is a randomized controlled trial that will be conducted at the American University of Beirut Medical Center - Delivery Suite.

DETAILED DESCRIPTION:
Women allocated to either the massage or compression group will be given 10 units of oxytocin intramuscularly immediately after delivery of the shoulder and controlled cord traction will be performed to assist placental delivery. The umbilical cord will be clamped and cut approximately 1 minute after delivery of the baby. The uterine fundus will be rubbed and blood clots expelled as quickly as possible after delivery of the placenta.

ELIGIBILITY:
Inclusion Criteria:

* Women giving birth vaginally, aged between 20 and 40 years, with a singleton pregnancy, gestational age of 36 or more weeks, and with fewer than or equal to three previous childbirths.

Exclusion Criteria:

* Exclusion criteria include multiple gestation, fetal malpresentation, the third stage of labor lasting more than 30 minutes, a previous cesarean delivery, chorioamnionitis, three or more previous induced abortions, preeclampsia, fetal death, polyhydramnios, hemoglobin of 9 g/L or less before delivery, coagulopathy, on magnesium sulfate infusion, abruptio placentae and having an abdominal wall too thick to palpate the fundus of the uterus or to perform uterine massage or compressions after delivery.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 445 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Incidence of blood loss of 500 mL or more | 2 years
  Collection of lost blood will be initiated immediately after delivery of the neonate by putting a drape under the woman's buttocks. Blood collected will be weighed on an electronic scale together with the drape, and the amount will be recorded in grams after subtracting the weight of the drape. The amount of blood loss will be recorded 30 mins after delivery of the neonate. The amount of lost blood in grams will be converted to volume by dividing by 1.06 (blood density in g/mL) for the analysis.

SECONDARY OUTCOMES:
Maternal pain | 2 years
  Maternal discomfort and pain intensity will be evaluated after the intervention using a visual analogue scale (VAS), which consists of a two-sided rule with a 10 cm vertical or horizontal line linking two points, at one extreme indicating a total absence of pain and at the other the worst pain imaginable. The women will be required to mark a spot on the line corresponding to the intensity of their pain at that particular time on a possible scale of 0 to 10.
Change in hemoglobin as a measure of blood loss | 2 years
  The change in hemoglobin will be defined as the mean difference of pre-delivery hemoglobin versus post-delivery hemoglobin in each group.
Use of therapeutic uterotonics | 2 years
  the need to use uterotonic agent for PPH such a misoprostol or ergotamines
Use of balloon or surgical procedures for postpartum hemorrhage | 2 years
  needingto insert tamponading devices such as balloon
Need for blood transfusion and hospital stay | 2 years
  needing to transfuse the patient due to severe anemia

CONTACTS AND LOCATIONS:
Overall Officials: Labib M Ghulmiyyah, MD, Principal Investigator — AUBMC
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Derived] Ghulmiyyah LM, El-Husheimi A, Usta IM, Colon-Aponte C, Ghazeeri G, Hobeika E, Mirza FG, Tamim H, Hamadeh C, Nassar AH. Effect of Sustained Uterine Compression versus Uterine Massage on Blood Loss after Vaginal Delivery: A Randomized Controlled Trial. Am J Perinatol. 2023 Nov;40(15):1644-1650. doi: 10.1055/s-0041-1739409. Epub 2021 Nov 14. PMID 34775581